CLINICAL TRIAL: NCT06759285
Title: Effect of Cradle Position on Comfort, Physiological Parameters and Vomiting Frequency in Premature Neonates During Orogastric Tube Feeding: A Randomized Controlled Trial
Brief Title: Effect of Cradle Position During Orogastric Tube Feeding on Comfort, Physiological Parameters and Vomiting
Acronym: CRADLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/89
Record Dates: First submitted 2024-12-22; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Position Differences; Nutrition; Nursing Care
Keywords: Preterm; Nutrition; Cradle position; Comfort; Vital signs; vomiting
MeSH Terms: conditions — Premature Birth; Vomiting

STUDY DESIGN:
Intervention Model Description: According to the sample size calculation made with G power 3.1.9.7, it was determined that 42 newborns (Experiment = 21, Control = 21) would meet the required sample size (0.96 effect size, 0.85 power, 0.05 margin of error). It was planned to include 24 newborns in each group, considering that there may be data losses. Since it was stated in the studies that it could affect gastric residue, randomization was performed by stratifying the feeding method. In order to ensure equal distribution in terms of nutrition in each group, two layers were created as breast milk and formula milk. The block/permutation method, which is one of the randomized assignment methods, was also used in the study. With this method, blocks containing equal numbers of A and B, symbolizing the experimental and control groups, were created using permutation and these blocks were multiplied until the specified number of people were reached. www.random.org was used to select the A and B block combination.
Who Masked: Participant
Masking Description: In the study, since the researcher was a clinical nurse who fed the babies and also carried out the data collection process, researcher blinding could not be done. However, babies were considered blind by nature. The analysis of the study was carried out by an independent statistician, the data were coded as A and B by coding the groups in the SPSS program, and statistical blinding was performed by not sharing the groups represented by the letters with the statistician to prevent bias. The stages of the study were carried out under the guidance of the Consolidated Standards of Reporting Trials (CONSORT) guide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cradle position (Experimental): The newborns in this group were swaddled and fed by being held in a cradle position on the nurse's lap during orogastric tube feeding.
  Interventions: Behavioral: Experimental (cradle position)
- Control Group (No Intervention): The newborns in this group were fed with an orogastric tube, in the supine position on a flat bed, with the head elevated, as is routine practice.

INTERVENTIONS:
Behavioral: Experimental (cradle position) — The newborn in cot bed was swaddled freely with the help of a thin blanket during feeding. Then, the nurse, wearing a box apron, took the baby in her arms and gave it a cradle position. The baby's physiological parameters and Comfort Scale were filled in before feeding began. The baby was kept in a cradle position on the researcher's lap during feeding. Immediately after feeding, without changing the baby's position, the physiological parameters and Comfort Scale were evaluated a second time, and again 15 minutes after feeding, without changing the position, the physiological parameters and Comfort Scale were evaluated a third time and recorded. Then, the baby was gently and slowly laid down on the denim bed as usual (right lateral).
  Arms: Cradle position

SUMMARY:
The study was planned to determine the effect of the cradle position applied during orogastric tube feeding in premature newborns on comfort, physiological parameters and vomiting frequency.

Hypotheses of the Study H1: The cradle position applied to premature newborns during orogastric tube feeding; H1a: It affects the comfort level compared to the control group. H1b: It affects physiological parameters compared to the control group. H1c: It affects the vomiting frequency compared to the control group.

DETAILED DESCRIPTION:
It is reported that the cradle position is the most preferred position by mothers during the breastfeeding process. The cradle position is a position where the mother holds the baby in her arms, the baby's head is placed on the inside of the mother's arm-elbow area, the baby's whole body is turned towards the mother, the baby's head is in line with the mother's breast, and the mother and the baby are in intense interaction. Although it is the most preferred position for breastfeeding, no study has been found in the literature evaluating the effect of the cradle position given during OGT feeding on the comfort level, physiological parameters and vomiting frequency of premature babies. For this reason, it is thought that it can be a supportive position that can be used by both neonatal nurses and mothers who are with their babies during the OGT feeding process for newborns preparing for the breastfeeding process in NICUs. It is thought that the study results will guide health workers and researchers regarding the supportive positions that should be given during newborn feeding.

ELIGIBILITY:
Inclusion Criteria:

* Having a feeding frequency of every 3 hours,
* Having a birth weight of 1000 grams and above,
* Having an indication for intermittent feeding (bolus) with OGT,
* Being placed in a bed,
* Not having a condition that prevents giving the cradle position (having undergone surgery, having a congenital anomaly, etc.)
* Having stable physiological parameters,
* Babies whose mothers were not with them during feeding (having undergone surgery, receiving inpatient treatment, being discharged and out of town, not wanting to be held during feeding, etc.) were included in the study.

Exclusion Criteria:

* • Continuous infusion, slow bolus feeding or parenteral nutrition method used for feeding,

  * Switching to full oral feeding,
  * Having nasal obstruction,
  * Receiving oxygen therapy, mechanical ventilation/CPAP support during the study period,
  * Receiving medication affecting gastrointestinal function during the study period (drugs that increase gastrointestinal tract motility and facilitate gastric emptying and gastrointestinal passage of nutrients, and drugs that decrease gastrointestinal tract motility).
  * Any medical diagnosis determined other than prematurity (Congenital anomaly, metabolic disease, asphyxia, sepsis, hyperbilirubinemia, intracranial hemorrhage and gastrointestinal hemorrhage, anatomic gastrointestinal anomaly, gastrointestinal disease, infection, frequent vomiting, distension).

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Newborn Information Form | First measurement:After admission in NICU 30th minutes
  This form was created by the researcher in accordance with the literature. The baby's gender, gestational week, birth weight, 1st and 5th APGAR Scores, postnatal day of study, corrected week, weight, amount of food and type of food were questioned.
Physiological Parameter Follow-up Form (Heart rate-min) | First feeding first measurement: 1 min before feeding
  The heart rate was measured after the baby was picked up and placed in the cradle position, just before orogastric tube feeding.
Physiological Parameter Follow-up Form (Respiration rate- min) | First feeding first measurement: 1 min before feeding
  Respiration rate was measured after the baby was picked up and placed in the cradle position, just before orogastric tube feeding.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | First feeding first measurement: 1 min before feeding
  Oxygen saturation was measured after the baby was picked up and placed in the cradle position, just before orogastric tube feeding.
Vomiting frequency tracking form | First feeding first measurement: 1 min before feeding
  The frequency of the baby's vomiting was recorded.
Stool amount tracking form | First feeding first measurement: 1 min before feeding
  The baby's stool volume was recorded.
Physiological Parameter Follow-up Form (Body temperature- 0C) | First feeding first measurement: 1 min before feeding
  Body temperature was measured after the baby was picked up and placed in the cradle position, just before orogastric tube feeding.
Abdominal Circumference Follow-up Form | First feeding first measurement: 1 min before feeding
  Abdominal circumference was measured while the baby was in bed, before the first feeding, and just before the nurse picked her/his up.
Neonatal Comfort Behavior Scale | First feeding first measurement: 1 min before feeding
  The first measurement was taken after the baby was picked up and just before starting to feed.

SECONDARY OUTCOMES:
Physiological Parameter Follow-up Form (Heart rate-min) | First feeding second measurement: 1 min after feeding
  The heart rate was measured a second time immediately after feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Respiration rate- min) | First feeding second measurement: 1 min after feeding
  Respiration rate was measured a second time immediately after feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | First feeding second measurement: 1 min after feeding
  Oxygen saturation was measured a second time immediately after feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Body temperature- 0C) | First feeding second measurement: 1 min after feeding
  Body temperature was measured a second time immediately after feeding while the baby was in the cradle position in the nurse's arms.
Neonatal Comfort Behavior Scale | First feeding second measurement: 1 min after feeding
  The second measurement was taken immediately after feeding with the baby in the cradle position.
Physiological Parameter Follow-up Form (Heart rate-min) | First feeding third measurement: 15 min after feeding
  The heart rate was measured for the third time at 15 minutes after feeding, while the baby was in the nurse's arms in the cradle position.
Physiological Parameter Follow-up Form (Respiration rate- min) | First feeding third measurement: 15 min after feeding
  Respiration rate was measured for the third time at 15 minutes after feeding, while the baby was in the nurse's arms in the cradle position.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | First feeding third measurement: 15 min after feeding
  Oxygen saturation was measured for the third time at 15 minutes after feeding, while the baby was in the nurse's arms in the cradle position.
Physiological Parameter Follow-up Form (Body temperature- 0C) | First feeding third measurement: 15 min after feeding
  Body temperature was measured for the third time at 15 minutes after feeding, while the baby was in the nurse's arms in the cradle position.
Neonatal Comfort Behavior Scale | First feeding third measurement: 15 min after feeding
  The third measurement was taken 15 minutes after feeding, with the baby in the cradle position on the nurse's lap.
Physiological Parameter Follow-up Form (Heart rate-min) | Second feeding first measurement: 1 min before feeding
  The heart rate was measured immediately before orogastric tube feeding after the baby was held in the cradle position.
Physiological Parameter Follow-up Form (Respiration rate- min) | Second feeding first measurement: 1 min before feeding
  Respiration rate was measured immediately before orogastric tube feeding after the baby was held in the cradle position.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Second feeding first measurement: 1 min before feeding
  Oxygen saturation was measured immediately before orogastric tube feeding after the baby was held in the cradle position.
Physiological Parameter Follow-up Form (Body temperature- 0C) | Second feeding first measurement: 1 min before feeding
  Body temperature was measured immediately before orogastric tube feeding after the baby was held in the cradle position.
Vomiting frequency tracking form | Second feeding first measurement: 1 min before feeding
  The frequency of the baby's vomiting was recorded.
Stool amount tracking form | Second feeding first measurement: 1 min before feeding
  The baby's stool volume was recorded.
Abdominal Circumference Follow-up Form | Second feeding first measurement: 1 min before feeding
  Abdominal circumference was measured while the baby was in bed, before the second feeding, and just before the nurse picked her/his up.
Neonatal Comfort Behavior Scale | Second feeding first measurement: 1 min before feeding
  The measurement was taken after the baby was picked up and just before starting to feed.
Physiological Parameter Follow-up Form (Heart rate-min) | Second feeding second measurement: 1 min after feeding
  The heart rate was measured a second time immediately after feeding in the second feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Respiration rate- min) | Second feeding second measurement: 1 min after feeding
  Respiration rate was measured a second time immediately after feeding in the second feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Second feeding second measurement: 1 min after feeding
  Oxygen saturation was measured a second time immediately after feeding in the second feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Body temperature- 0C) | Second feeding second measurement: 1 min after feeding
  Body temperature was measured a second time immediately after feeding in the second feeding while the baby was in the cradle position in the nurse's arms.
Neonatal Comfort Behavior Scale | Second feeding second measurement: 1 min after feeding
  The second measurement was taken immediately after feeding with the baby in the cradle position in the second feeding.
Physiological Parameter Follow-up Form (Heart rate-min) | Second feeding third measurement: 15 min after feeding
  The heart rate was measured third time immediately after feeding in the second feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Respiration rate- min) | Second feeding third measurement: 15 min after feeding
  was measured third time immediately after feeding in the second feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Second feeding third measurement: 15 min after feeding
  Respiration rate was measured third time immediately after feeding in the second feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Body temperature- 0C) | Second feeding third measurement: 15 min after feeding
  Body temperature was measured third time immediately after feeding in the second feeding while the baby was in the cradle position in the nurse's arms.
Neonatal Comfort Behavior Scale | Second feeding third measurement: 15 min after feeding
  The third measurement was taken immediately after feeding with the baby in the cradle position in the second feeding.
Physiological Parameter Follow-up Form (Heart rate-min) | Third feeding first measurement: 1 min before feeding
  Heart rate was measured first time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Respiration rate- min) | Third feeding first measurement: 1 min before feeding
  Respiration rate was measured first time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Third feeding first measurement: 1 min before feeding
  Oxygen saturation was measured first time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Body temperature- 0C) | Third feeding first measurement: 1 min before feeding
  Body temperature was measured first time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Vomiting frequency tracking form | Third feeding first measurement: 1 min before feeding
  The frequency of the baby's vomiting was recorded.
Stool amount tracking form | Third feeding first measurement: 1 min before feeding
  The baby's stool volume was recorded.
Abdominal Circumference Follow-up Form | Third feeding first measurement: 1 min before feeding
  Abdominal circumference was measured while the baby was in bed, before the third feeding, and just before being picked up by the nurse.
Neonatal Comfort Behavior Scale | Third feeding first measurement: 1 min before feeding
  The first measurement was taken immediately after the third feeding with the baby in the cradle position in the second feeding.
Physiological Parameter Follow-up Form (Heart rate-min) | Third feeding second measurement: 1 min after feeding
  Heart rate was measured second time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Respiration rate- min) | Third feeding second measurement: 1 min after feeding
  Respiration rate was measured second time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Third feeding second measurement: 1 min after feeding
  Oxygen saturation was measured second time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Body temperature- 0C) | Third feeding second measurement: 1 min after feeding
  Body temperature was measured second time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Neonatal Comfort Behavior Scale | Third feeding second measurement: 1 min after feeding
  The second measurement was taken immediately after the third feeding with the baby in the cradle position in the second feeding.
Physiological Parameter Follow-up Form (Heart rate-min) | Third feeding third measurement: 15 min after feeding
  Heart rate was measured third time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Respiration rate- min) | Third feeding third measurement: 15 min after feeding
  was measured third time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Oxygen saturation -SpO2%) | Third feeding third measurement: 15 min after feeding
  Respiration rate was measured third time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Physiological Parameter Follow-up Form (Body temperature- 0C) | Third feeding third measurement: 15 min after feeding
  Body temperature was measured third time immediately after third feeding while the baby was in the cradle position in the nurse's arms.
Neonatal Comfort Behavior Scale | Third feeding third measurement: 15 min after feeding
  The third measurement was taken immediately after the third feeding with the baby in the cradle position in the second feeding.

CONTACTS AND LOCATIONS:
Overall Officials: sibel küçükoğlu, Prof, Study Director — Selcuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Sibel Küçükoğlu, Selçuklu, Akademi Mahallesi
  - Sibel Kucukoglu, Konya

IPD SHARING:
Plan to Share IPD: No